CLINICAL TRIAL: NCT03350308
Title: Prediction of Risk of Hypotension in Hemodialysis
Acronym: IMHOTEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fresenius Medical Care North America (Industry); Centre de dialyse AURA Plaisance (Unknown); Pôle Santé République (Other); Service de Néphrologie et Hémodialyse (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-363; 2014-A01538-39 (Other: 2014-A01538-39-+)
Record Dates: First submitted 2017-11-15; First posted 2017-11-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Chronical Kidney Disease; Hypotension; Residual Blood Volume; Hemodialysis
MeSH Terms: conditions — Hypotension | interventions — Renal Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic end-stage renal failure
  Interventions: Other: hemodialysis

INTERVENTIONS:
Other: hemodialysis — The main objective is to establish a statistical predictive model of the risk of intradialytic hypotension during hemodialysis (HD) or hemodiafiltration (HDF) sessions based on the measurement of residual blood volume and excess extracellular hydration

SUMMARY:
The main objective is to establish a statistical predictive model of the risk of intradialytic hypotension during hemodialysis (HD) or hemodiafiltration (HDF) sessions based on the measurement of residual blood volume and excess extracellular hydration. The secondary objective is to study the impact of dysfunction in the mechanisms of compensation for decreased blood volume (heart disease, neuropathy, drugs) on the risk of intradialytic hypotension.

DETAILED DESCRIPTION:
The duration of the study is 4 weeks for each patient. It will first be carried out a spectral analysis of heart rate variability (CHU of Clermont Ferrand only) and a measurement of intracellular and extracellular volumes by bioimpedancemetry. During the next 9 sessions, the decrease in the VSR will be recorded using an optical haematocrit measurement system. Blood pressure and heart rate will be measured every 30 minutes using an automatic blood pressure monitor and whenever the patient's nurse deems it necessary.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old minimum patients
* Patients with chronic end-stage renal failure
* Patients treated with hemodialysis for at least 3 months, 3 times a week (duration of sessions 3 to 5 hours)
* Patients with at least 2 episodes of intradialytic hypotension in the last month
* Patients without acute events within 3 months prior to inclusion
* Patients affiliated with or receiving social security benefits

Exclusion Criteria:

* Hemoglobin levels outside the limits of measurement (<7 g/L or >15g/L)
* Patients whose probable survival does not exceed 6 months
* Patients with progressive acute pathology
* Patient following another research protocol that may influence results
* Patients with psychiatric pathology or cognitive impairments that make them unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic end-stage renal failure
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Risk of PAS with symptom | at 3 week
  The primary outcome will be the risk of a decrease in PAS of more than 20 mmHg or a decrease in WFP of at least 10 mmHg associated with clinical symptomatology (vertigo, malaise, nausea or cramps)

SECONDARY OUTCOMES:
Risk of PAS with symptom without symptom | at 3 week
  The risk of a decrease in PAS of more than 20 mmHg or a decrease in WFP of at least 10 mmHg (with or without symptoms)
risk of reduction of PAS below 90 mmHg (with or without symptoms) | at 3 week
risk of isolated symptoms caracterized by vertigo, discomfort, nausea or cramps | at 3 week

CONTACTS AND LOCATIONS:
Overall Officials: Julien ANIORT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France